CLINICAL TRIAL: NCT00859872
Title: Efficacy and Safety of Risperidone Oral Solution Combination Clonazepam Versus Haloperidol IM Injection for Treatment of Acute Psychotic Agitation in Schizophrenia
Brief Title: Efficacy and Safety of Risperidone Oral Solution Combination Clonazepam Versus Haloperidol Intramuscular (IM) Injection for Treatment of Acute Psychotic Agitation in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central South University (Other)
Collaborators: Wuhan Mental Health Institute (Unknown); Capital Medical University (Other); Shanghai Mental Health Center (Other); Guangzhou Mental Hospital (Other); Chongqing Mental Hospital (Unknown)
Responsible Party: MentalHealth Institute of the 2nd Xiangya Hospital, Central South University, the 2nd Xiangya Hospital, Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIS-0801
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Schizophrenia
Keywords: acute psychotic agitation; schizophrenia; risperidone oral solution; clonazepam; haloperidol
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Haloperidol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral group (Experimental): risperidone oral solution combination clonazepam oral
  Interventions: Drug: risperidone oral solution
- IM group (Active Comparator): haloperidol IM injection
  Interventions: Drug: haloperidol

INTERVENTIONS:
Drug: risperidone oral solution — risperidone oral solution (2-6mg/d) combination clonazepam (4-8mg/d) oral
  Arms: oral group
Drug: haloperidol — haloperidol IM injection (5-20mg/d)
  Arms: IM group

SUMMARY:
This is a multi-centre, open, randomized, haloperidol-referenced, 47 days two treatment sessions, parallel-group study.

After screening period, eligible subjects will be entered 5 days treatment session I to compare the efficacy between risperidone oral solution combination clonazepam oral and haloperidol IM injection on controlling psychotic agitation, then will be followed by 6 additional weeks treatment session II for exploring the effect of medicine switching from IM injection to oral.

DETAILED DESCRIPTION:
Acute psychotic agitation is a common problem in many patients with schizophrenia that includes agitation, aggression, excitement and violence. An investigation showed that about 26% psychotic patients were brought to the psychiatric emergency room because of the psychotic agitation symptoms. The primary objective is to compare the efficacy between risperidone oral solution combination clonazepam oral and haloperidol IM injection on controlling psychotic agitation in patients of acute schizophrenia and schizophrenic-affective disorder.

The secondary objectives are: (1) to explore the possibility of decreasing efficacy of acute 6 weeks treatment from IM injection to oral; (2) to compare the safety between risperidone oral solution combination clonazepam oral and haloperidol IM injection.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 45 years
* DSM-IV diagnosis of acute exacerbation of schizophrenia or schizoaffective disorders
* A score of ≥ 14 on a 5-item acute-agitation cluster (including excitement, hostility, uncooperativeness and poor impulse control) derived from the PNASS
* The total scores ≥60 on the PANSS

Exclusion Criteria:

* Women who are pregnant or breast feeding, or who plan to become pregnant during the study
* The psychotic agitation is caused by delirium, epilepsy, mental retardation and affective disorder; intoxication or symptoms of withdrawal from alcohol or other psychoactive substances
* Clinical laboratory values indicating serious medical illness
* Known hypersensitivity to any of the study medications
* Treatment with a depot antipsychotic with 1 cycle of screening
* Using of disallowed medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
the change of PANSS-EC scores | 5 days

SECONDARY OUTCOMES:
response rate based on the PANSS | 47 days

CONTACTS AND LOCATIONS:
Locations (1):
- MentalHealth Institute of the 2nd Xiangya Hospital, Central South University, Changsha, Hunan, China